CLINICAL TRIAL: NCT06939153
Title: Effects of Age, Sex and Isometric Exercise on Ventricular-Vascular Interactions During Cardiac Unloading
Acronym: Unload heart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tracy Baynard (Other)
Responsible Party: Sponsor-Investigator, Tracy Baynard, Professor/Associate Vice Provost for Graduate Education, University of Massachusetts, Boston
Organization: University of Massachusetts, Boston (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 4001
Record Dates: First submitted 2025-03-28; First posted 2025-04-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Orthostatic Intolerance
MeSH Terms: conditions — Orthostatic Intolerance | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Young male adults (Active Comparator): All young males will complete both conditions under study: 1) LBNP and LBNP + isometric handgrip exercise
  Interventions: Other: LBNP; Other: LBNP + Isometric handgrip exercise
- Young females (Active Comparator): All young females will complete both conditions under study: 1) LBNP and LBNP + isometric handgrip exercise
  Interventions: Other: LBNP; Other: LBNP + Isometric handgrip exercise
- Older male adults (Active Comparator): All older males will complete both conditions under study: 1) LBNP and LBNP + isometric handgrip exercise
  Interventions: Other: LBNP; Other: LBNP + Isometric handgrip exercise
- Older female adults (Active Comparator): All older females will complete both conditions under study: 1) LBNP and LBNP + isometric handgrip exercise
  Interventions: Other: LBNP; Other: LBNP + Isometric handgrip exercise

INTERVENTIONS:
Other: LBNP — Participants will be exposed to a lower body negative pressure chamber protocol consisting of 5-min stages in the order of 20, -30, -40 and -50 mmHg.
Other: LBNP + Isometric handgrip exercise — Participants will undergo 5-minute stages of LBNP at -20, -30, -40, and -50 mmHg in sequence. During the -30, -40, and -50 mmHg stages, they will perform a 2-minute isometric handgrip exercise, starting at the third minute and sustaining it for the remaining duration.

SUMMARY:
As people get older, especially women, they often feel dizzy or even faint when they go from sitting or lying down to standing up. This happens because their blood pressure (BP) drops, which can lead to falls, heart problems, and even death in older adults. When BP changes, it affects how well the heart works and how it talks with blood vessels. However, little research has been done on how the heart and blood vessels talk during times of low BP. The crosstalk between the heart and blood vessels is important, as it allows enough blood and oxygen to reach the brain and other vital organs. Some research shows that as we get older, the crosstalk does not work as well. This can make it harder for blood to flow properly or put extra pressure on the heart and arteries. That's why we want to study how the heart and blood vessels talk during a laboratory-simulated situation of low BP in young and older men and women. In our study, participants will lie down with their lower body in a chamber that creates a vacuum around their legs. This safely mimics what happens when you stand up quickly. We can then measure heart function, the stress on arteries, and BP while your legs are in that vacuum. We'll use an ultrasound to check the heart and a finger cuff to measure BP. We'll also see if gripping something firmly can help protect from sudden drops in blood pressure. This study will help us understand more about a condition called orthostatic hypotension and might even suggest that handgrip exercise could prevent it.

The main questions the current study aims to address are:

* Does the cross-talk between the heart and vessels become more impaired with aging during laboratory-simulated conditions of low BP?
* Do women have worse crosstalk between the heart and blood vessels during laboratory-simulated conditions of BP?
* Does hand gripping protect against drops in BP during conditions of low BP?

All participants will be asked to

* Complete two laboratory conditions on two separate days with a randomized order (like flipping a coin):
* Exposure to a lower body negative pressure (LBNP) chamber to safely simulate low BP (control)
* Exposure to a lower body negative pressure (LBNP) while conducting hand-squeezingexercise (experimental).

The investigators will examine how heart and blood vessel interactions, as well as blood pressure (BP) responses, differ in young and older adults of both sexes when exposed to a laboratory-simulated low BP condition (LBNP), both with and without hand squeezing exercise.

DETAILED DESCRIPTION:
Orthostatic intolerance becomes prevalent with advancing age (≤5% below age 50 but ~20% above age 70), and females are 3 to 5% more susceptible. Orthostatic intolerance is associated with syncope, falls, cardiovascular disease, and mortality in older adulthood. The characteristic excessive fall in blood pressure (BP) underlies a complex dysregulation of heart rate (HR), BP, and flow responses to postural changes. When standing, blood pools in the lower limbs, decreasing venous return, stroke volume (SV), and ultimately BP. The resultant unloading of the heart upregulates the sympathetic arm of the baroreflex to increase HR and peripheral vasoconstriction, but this counter-regulation to restore normal BP appears absent or reduced in people suffering from orthostatic intolerance.

Cardiac unloading, which can be accomplished experimentally via lower body negative pressure (LBNP), produces changes in arterial and ventricular loads while attempting to maintain adequate cardiac output. Heart-vessel interactions are, thus, key to understanding BP regulation during cardiac unloading, but have been ignored by research on orthostatic intolerance. The ventricular-vascular coupling framework based on pressure-volume loops describes how heart contractility (i.e., ventricular elastance (Ees)) and arterial loads (i.e., arterial elastance (Ea)), respond to changing loading conditions. With aging, females show greater increases in Ees to match increased Ea, caused by aortic stiffening and high BP. Hence, the coupling ratio (Ea/Ees) is reduced in females, but is preserved in males. However, whether such changes at rest impact the ventricular-vascular coupling response to acute cardiac unloading is unknown, and may be an important mechanism of orthostatic intolerance in females. Notably, the ventricular-vascular coupling framework disregards the wave reflection phenomenon underlying pulsatile pressure-flow relationships. Early reflection of pressure waves, which is characteristic of aging, increases cardiac afterload and thus has important implications for heart-vessel interactions. Such pulsatile arterial load is expected to rise in response to cardiac unloading due to peripheral vasoconstriction, but this remains untested. Importantly, defining heart-vessel interactions during cardiac unloading will shed light on whether plausible ventricular-vascular mismatch contributes to orthostatic intolerance and may help to develop countermeasures to alleviate the symptoms and consequences of intolerance.

Isometric exercise attenuates the cardiac unloading effects via increases in both cardiac output and BP. The pressor response elicited by isometric handgrip exercise increases both heart and arterial load. While isometric handgrip exercise holds potential to counteract BP reduction during cardiac unloading, the augmented work of the heart may limit tolerance. Thus, defining the effects of isometric handgrip exercise on ventricular-vascular interactions under cardiac unloading and the impact of age and sex on these responses will be key to determining its feasibility as an orthostatic intolerance countermeasure.

Therefore, our specific aims are to determine the impact of age (Aim 1), sex (Aim 2), and isometric handgrip exercise (Aim 3) on ventricular-vascular interactions during LBNP-induced cardiac unloading.

* Aim 1's working hypothesis is that older, compared to young healthy adults will exhibit a more pronounced ventricular-vascular mismatch due to greater increases in Ea and Ew not matched by Ees during presyncope- limited LBNP.
* Aim 2's working hypothesis is that older but not younger healthy females compared to males will exhibit a more pronounced ventricular-vascular mismatch due to smaller increases in Ea and Ew and higher Ees during presyncope-limited LBNP.
* Aim 3's working hypothesis is that isometric handgrip exercise will offset BP reductions, but increase ventricular and arterial load during presyncope- limited LBNP.

ELIGIBILITY:
Inclusion Criteria

* People aged 18-35 years or aged ≥ 65 years
* Healthy without symptons of orthostatic intolerance (i.e., nausea, sweating, weakness, visual disturbance)
* Seated systolic and/or diastolic BP <140/90 mmHg;
* Body mass index <35 kg/m2
* Recreationally active (≤ 2 days of structured physical activity)
* Regular menstrual cycles in young females

Exclusion Criteria:

* People diagnosed with cardiovascular, diabetes, inflammatory or renal diseases and neurodegenerative-related dementia
* Tobacco users
* People prescribed with beta-blockers
* Pregnant females
* People unable to fit or get into the lower body negative pressure chamber

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Arterial elastance | "Baseline/pre-LBNP", "During each LBNP stage (-20 mmHg, -30 mmHg, -40 mmHg, -50 mmHg) in the last 2 minutes"
  Arterial elastance reflective of lumped afterload will be non-invasively estimated as end-systolic pressure (obtained from tonometry) divided by stroke volume (obtained from echocardiography)
Ventricular elastance | "Baseline/pre-LBNP", "During each LBNP stage (-20 mmHg, -30 mmHg, -40 mmHg, -50 mmHg) in the last 2 minutes"
  Ventricular elastance, reflective of ventricle contractility, will be non-invasively estimated as end-systolic pressure (obtained from tonometry) divided by end-systolic volume (obtained from echocardiography).
Ventricular-vascular coupling ratio | "Baseline/pre-LBNP", "During each LBNP stage (-20 mmHg, -30 mmHg, -40 mmHg, -50 mmHg) in the last 2 minutes"
  The arterial-to-ventricular elastance ratio will be considered as an index describing cardiac energy and efficacy.
Wasted pressure effort | "Baseline/pre-LBNP", "During each LBNP stage (-20 mmHg, -30 mmHg, -40 mmHg, -50 mmHg) in the last 2 minutes"
  Wasted pressure effort, a marker of pulsatile afterload, will be estimated from pressure-flow analyses
Brachial blood pressure | "Baseline/pre-LBNP", "During each LBNP stage (-20 mmHg, -30 mmHg, -40 mmHg, -50 mmHg) in the last 2 minutes"
  Beat-to-beat BP will be recorded continuously using finger plethysmography and calibrated to reflect both brachial artery systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained in this study may be provided to qualified researchers with an academic interest in orthostatic intolerance. Data or samples shared will be coded, with no personal health information included. Approval of the request and execution of all applicable agreements (i.e., a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.

REFERENCES:
- [Background] Stock JM, Shenouda N, Chouramanis NV, Patik JC, Martens CR, Farquhar WB, Chirinos JA, Edwards DG. Effect of acute handgrip and aerobic exercise on wasted pressure effort and arterial wave reflections in healthy aging. Am J Physiol Heart Circ Physiol. 2023 Oct 1;325(4):H617-H628. doi: 10.1152/ajpheart.00133.2023. Epub 2023 Jul 21. PMID 37477688
- [Background] Stratton JR, Halter JB, Hallstrom AP, Caldwell JH, Ritchie JL. Comparative plasma catecholamine and hemodynamic responses to handgrip, cold pressor and supine bicycle exercise testing in normal subjects. J Am Coll Cardiol. 1983 Jul;2(1):93-104. doi: 10.1016/s0735-1097(83)80381-7. PMID 6853921
- [Background] Goswami N, Blaber AP, Hinghofer-Szalkay H, Convertino VA. Lower Body Negative Pressure: Physiological Effects, Applications, and Implementation. Physiol Rev. 2019 Jan 1;99(1):807-851. doi: 10.1152/physrev.00006.2018. PMID 30540225
- [Background] Ricci F, Fedorowski A, Radico F, Romanello M, Tatasciore A, Di Nicola M, Zimarino M, De Caterina R. Cardiovascular morbidity and mortality related to orthostatic hypotension: a meta-analysis of prospective observational studies. Eur Heart J. 2015 Jul 1;36(25):1609-17. doi: 10.1093/eurheartj/ehv093. Epub 2015 Apr 6. PMID 25852216
- [Background] Fu Q, Arbab-Zadeh A, Perhonen MA, Zhang R, Zuckerman JH, Levine BD. Hemodynamics of orthostatic intolerance: implications for gender differences. Am J Physiol Heart Circ Physiol. 2004 Jan;286(1):H449-57. doi: 10.1152/ajpheart.00735.2002. Epub 2003 Oct 2. PMID 14527942
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Fedorowski A, Ricci F, Hamrefors V, Sandau KE, Hwan Chung T, Muldowney JAS, Gopinathannair R, Olshansky B. Orthostatic Hypotension: Management of a Complex, But Common, Medical Problem. Circ Arrhythm Electrophysiol. 2022 Mar;15(3):e010573. doi: 10.1161/CIRCEP.121.010573. Epub 2022 Feb 25. PMID 35212554